CLINICAL TRIAL: NCT06160180
Title: Randomized Controlled Trial on Assessment of Preoperative Versus Postoperative Submucosal Dexamethasone On Postoperative Complications Following Surgical Extraction Of Mandibular Third Molar.
Brief Title: Comparative Assessment of Preoperative Versus Postoperative Submucosal Dexamethasone on Postoperative Complications Following Surgical Extraction of Mandibular Third Molar: Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Shristi Maharjan, Junior Resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRC/2508/023
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug arm preoperative (Active Comparator): Injection 2ml of 4mg dexamethasone loaded and deposited submucosally in the buccal vestibule of the extraction site after local anesthesia but before placement of the first incision.
  Interventions: Drug: Dexamethasone
- Drug arm postoperative (Active Comparator): Injection 2ml of 4mg dexamethasone loaded and deposited submucosallyin the buccal vestibule of the extraction site after finishing extraction and placement of last suture.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Submucosal application
  Other Names: treatment

SUMMARY:
The goal of this study is to compare the pain, edema and trismus of pre-operative versus post-operative submucosal dexamethasone in lower third molar surgical extraction done in healthy population.This is comparative study, will be conducted in patient indicated for surgical extraction of mandibular third molar at the department of oral and maxillofacial surgery, college of dental surgery, BPKIHS, Nepal. Verbal and written informed consent will be taken. Participants meeting inclusion criteria will be included in the study and will be divided into two groups, group A(pre-operative submucosal 2ml of 4mg/ml dexamethasone will be administered prior to placing an incision in buccal vestibule) and groupB(post-operative submucosal 2ml of 4mg/ml dexamethasone will be administered soon after closure of the incision site).Baseline measurement of interincisal distance for mouth opening, distance between the tragus to corner of mouth, gonion to corner of mouth and outer canthus to gonion as baseline for edema taken prior extraction. Extraction is carried out using standard protocol and postoperative antibiotics and analgesics are given. Rescue analgesic tramadol is prescribed and asked to be taken only pain score exceeds 7.Patient is kept on follow up for 2nd, 5th and 7th days and assessment of pain using numeric visual analogue scale, swelling using facial and trismus using interincial measurements and recorded. Any adverse effect of drugs will be recorded. The data collected will be entered in Microsoft excel sheet. It will then be transferred into SPSS(Statistical package for Social Sciences) for statistical analysis.

DETAILED DESCRIPTION:
Introduction:Third molar impaction is a chronic disorder that often necessitates tooth extraction. Impaction is characterized as the inability of a tooth to erupt at its proper location in the dental arch during its usual growth time.The surgical extraction of lower third molars is the most frequent intervention in oral surgery. This procedure is often associated with significant postsurgical sequelae that may have both biological and social impact. Besides severe complications such as dysaesthesia, severe infection, fracture, and dry socket, patients frequently complain of pain, swelling, and limitation in mouth opening (Trismus) throughout the postoperative course due to the inflammatory response following the surgical injury. To control postoperative inflammation and symptoms associated, it is necessary to provide an adequate anti-inflammatory therapy and various medications have been prescribed for the same. For several decades surgeons administered corticosteroids before or just after third molars' surgery to reduce inflammation and associated symptoms after oral surgery. Corticosteroids mechanism of action is the inhibition of the enzyme Phospholipase A2 (PLA 2), which reduces the release of arachidonic acid in the cells of the inflamed area.This will decrease prostaglandins and leukotriene synthesis; therefore reducing the accumulation of neutrophils has been the greatest advantage of corticosteroids compared to non-steroidal anti-inflammatory drugs. The aim of this study was to evaluate the effect of preoperative versus postoperative administration of submucosal Dexamethasone on postoperative discomfort including pain, edema, and trismus following lower third molar surgery in order to allow a better welfare of the patient and to return the patient to the normal activity following the surgery. And to determine the efficacy of single dose 2 ml/8 mg submucosal dexamethasone injection in the buccal vestibule in proximity to the surgical site.

Rational:Pain and edema are the most frequent postoperative sequelae to surgical removal of impacted teeth, all of which are due to the local inflammatory response. The inflammation induced by tissue damage is the primary cause of acute postoperative pain after third molar extraction. Edema after third molar surgery is caused by extravasation of fluid by traumatized tissues as a consequence of the disruption or obstruction of lymph arteries, culminating in the termination of lymph drainage, which accumulates in the tissues. Adjunctive use of corticosteroids to decrease tissue mediators of inflammation and reduce fluid transudation and edema is common in surgical procedures. Corticosteroids inhibits the enzyme Phospholipase A2 (PLA 2), which reduces the release of arachidonic acid in the cells of the inflamed area.Dexamethasone has higher potency, lower sodium retaining ability and longer half-life. Long-acting steroids outperform short-acting steroids, and submucosal steroid administration has similar consequences as intravenous and intramuscular routes. Also rate of absorption is highly dependent on the blood flow to the site.Submucosal dexamethasone is quite simple, less invasive, painless, convenient for the surgeon and the patient and offers a low cost solution for the typical discomfort associated with the extraction of impacted lower third molar. Also,submucosal injection offers advantage of concentrating the drug near the surgical area with less systemic absorption and no further manipulation of the tissues.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy patients (American Society of Anesthesiology I) with impacted lower third molar.
* Age ≥18 to ≤ 55 years
* No history of previous pericoronitis

Exclusion Criteria:

* • Patients who are ASA II to ASA VI.

  * Patients already on corticosteriods through any route.
  * Patients with known allergy to any drugs.
  * Pregnant and lactating females
  * Patient not consenting to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
PAIN MEASUREMENT POSTOPERATIVELY AFTER SURGICAL EXTRACTION OF 3RD MOLAR | SECOND, FIFTH AND SEVENTH POST OPERATIVE DAY
  Pain will be calculated through Visual analogue Scale with 1 being least painful and 10 being most painful. Each patient fter extraction will be instructed for follow up in 2nd 5th and 7th postoperative days and asked to give value for the pain they experienced.
  Number of analgesics consumed was also counted from 2nd postoperative day to 7th postoperative day and will be recorded in written logbook.
  Number of resucue analgesics: if in case of severe pain not relieved by prescribed analgesic(Tab paracetamol+ ibuprofen), Cap tramadol is prescribed if necessary and was recorded in each postoperative days and written in the log book.
SWELING | BASELINE,SECOND, FIFTH AND SEVENTH POSTOPERATIVE DAY
  facial measurements through graduated measuring tape in centimeters (outer canthus to gonion, tragus of ear to corner of mouth and corner of mouth to gonion
TRISMUS | BASELINE,SECOND, FIFTH AND SEVENTH POSTOPERATIVE DAY
  MEASURING NON-FORCED INTERINCISAL DISTANCE THROUGH STANDARD MEASURING SCALE IN MILIMETERS

REFERENCES:
- [Background] Lau AAL, De Silva RK, Thomson M, De Silva H, Tong D. Third Molar Surgery Outcomes: A Randomized Clinical Trial Comparing Submucosal and Intravenous Dexamethasone. J Oral Maxillofac Surg. 2021 Feb;79(2):295-304. doi: 10.1016/j.joms.2020.09.020. Epub 2020 Sep 17. PMID 33058774
- [Background] Saravanan K, Kannan R, John RR, Nantha Kumar C. A Single Pre Operative Dose of Sub Mucosal Dexamethasone is Effective in Improving Post Operative Quality of Life in the Surgical Management of Impacted Third Molars: A Comparative Randomised Prospective Study. J Maxillofac Oral Surg. 2016 Mar;15(1):67-71. doi: 10.1007/s12663-015-0795-0. Epub 2015 May 26. PMID 26929555
- [Background] Al-Shamiri HM, Shawky M, Hassanein N. Comparative Assessment of Preoperative versus Postoperative Dexamethasone on Postoperative Complications following Lower Third Molar Surgical Extraction. Int J Dent. 2017;2017:1350375. doi: 10.1155/2017/1350375. Epub 2017 Apr 10. PMID 28487738
- [Background] Deo SP. Effect of submucosal injection of dexamethasone on post-operative sequelae of third molar surgery. JNMA J Nepal Med Assoc. 2011 Apr-Jun;51(182):72-8. PMID 22916516
- [Background] Majid OW, Mahmood WK. Effect of submucosal and intramuscular dexamethasone on postoperative sequelae after third molar surgery: comparative study. Br J Oral Maxillofac Surg. 2011 Dec;49(8):647-52. doi: 10.1016/j.bjoms.2010.09.021. Epub 2010 Oct 29. PMID 21035237
- [Background] Bhargava D, Sreekumar K, Deshpande A. Effects of intra-space injection of Twin mix versus intraoral-submucosal, intramuscular, intravenous and per-oral administration of dexamethasone on post-operative sequelae after mandibular impacted third molar surgery: a preliminary clinical comparative study. Oral Maxillofac Surg. 2014 Sep;18(3):293-6. doi: 10.1007/s10006-013-0412-7. Epub 2013 Mar 20. PMID 23512235
- [Background] Almeida RAC, Lemos CAA, de Moraes SLD, Pellizzer EP, Vasconcelos BC. Efficacy of corticosteroids versus placebo in impacted third molar surgery: systematic review and meta-analysis of randomized controlled trials. Int J Oral Maxillofac Surg. 2019 Jan;48(1):118-131. doi: 10.1016/j.ijom.2018.05.023. Epub 2018 Jun 23. PMID 29941229